CLINICAL TRIAL: NCT04130269
Title: The Impact of Anxiety, Stress and Pain in the Early Phase of Myocardial Infarction on the Development of Anxiety Symptoms and Posttraumatic Stress Disorder in the Long Term Outcome
Brief Title: Anxiety, Stress and Pain & Myocardial Infarction
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 7479; 31-478 ex 18/19 (Other: Ethikkommission, Medical University of Graz)
Record Dates: First submitted 2019-10-16; First posted 2019-10-17 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with MCI: Patients with myocardial infarction (STEMI/NSTEMI) aged 19-90
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Questionnaires, lab-run

SUMMARY:
People often experience the acute phase of a myocardial infarction as a stressful and traumatic event that seems lifethreatening. Such anxiety, pain and stress can lead to the development of posttraumatic stress disorder in the long run. Previous studies suggest that there might be a relevant percentage of people developing Posttraumatic Stress Disorder (PTSD) after a myocardial infarction. Posttraumatic stress disorder is a risk factor for the development of coronary heart disease. The goal of this study is to detect the percentage of people that develop symptoms of anxiety, stress, and PTSD after an acute myocardial infarction.

DETAILED DESCRIPTION:
People often experience the acute phase of a myocardial infarction as a stressful and traumatic event that seems lifethreatening. Such anxiety, pain and stress can lead to the development of posttraumatic stress disorder in the long run. Previous studies suggest that there might be a relevant percentage of people developing PTSD after a myocardial infarction. Posttraumatic stress disorder is a risk factor for the development of coronary heart disease. The goal of this study is to detect the percentage of people that develop symptoms of anxiety, stress and PTSD after an acute myocardial infarction.

Patients will be examined during three times - in the acute myocardial infarction period (Day 1-3), before dismissal (Day 5-14) and after 6 months for a follow-up. During all times they will be given questionnaires asking about their levels of stress, anxiety and general well-being as well as tests checking their cognitive abilities (thus to find out if they decrease over time). Moreover, blood samples checking cortisol levels as well as metanephrine levels will be taken in order to objectify the levels of stress that are stated by the patients. Furthermore, clinical evaluations, laboratory runs (troponin), ECGs and echocardiographies will be done at all three points in time.

The goal is to detect the biopsychosocial relations and to develop better prevention.

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate in the study
* men and women 19-90
* after myocardial infarctions
* no psychiatric disease before myocardial infarction
* no other severe disease influencing the immune system

Exclusion Criteria:

* non fulfilment of inclusion criteria
* non-compliant patients (dementia, delirium)
* steroid-therapy

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women 19-90.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-07 (Actual); Primary Completion 2027-12-07 (Estimated); Study Completion 2027-12-07 (Estimated)

PRIMARY OUTCOMES:
PTSD | 6 months
  Number of patients who develop PTSD

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided